CLINICAL TRIAL: NCT00002950
Title: Phase I/II Study of Topotecan (SKF 104864) With Recombinant GM-CSF (Sargramostim) Used as a Priming Agent in Advanced Malignancies
Brief Title: Topotecan Plus Sargramostim in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065420; YALE-HIC-9043 (Other: Yale Human Investigations Committee); NCI-G97-1158 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-03-26 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — sargramostim; Topotecan

INTERVENTIONS:
Biological: sargramostim
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase I/II trial to study the effectiveness of topotecan plus sargramostim in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Identify a priming schedule of sargramostim (GM-CSF) that reduces the percentage of progenitor cells in cycle at the time of chemotherapy administration in patients with advanced malignancies. II. Determine the maximum tolerated dose and toxic effects of topotecan when administered with sargramostim in these patients. III. Conduct a preliminary assessment of the activity of this topotecan regimen in these patients.

OUTLINE: This is a dose escalation study of topotecan. Patients receive priming with sargramostim (GM-CSF) on days -4 through -2. On day 0, topotecan IV is administered over 30 minutes. Cohorts of 6 patients receive escalating doses of topotecan. The maximum tolerated dose (MTD) is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity (DLT). Sargramostim resumes on day 1 following topotecan, and continues for 5 days or until sufficient hematologic recovery. The next course of topotecan is given 48 hours later. Treatment repeats every 6 weeks for 4 courses. Patients are followed every 3 months for the first year, then every 6 months thereafter.

PROJECTED ACCRUAL: 15-25 patients will be accrued for the duration of 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven malignancy for which no alternative treatment exists

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Platelet count at least 100,000/mm3 Absolute neutrophil count at least 1500/mm3 Hepatic: Total bilirubin no greater than 2.0 mg/dL Renal: Creatinine clearance at least 50 mL/min Other: No active infections HIV negative No other concurrent medical condition

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) Endocrine therapy: Not specified Radiotherapy: No prior wide field radiotherapy No prior radiotherapy to greater than 20% of bone marrow Surgery: Recovered from prior surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1996-09-26 (Actual); Primary Completion 2002-02-10 (Actual); Study Completion 2002-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Rutherford, MD, PhD, Study Chair — Yale University
Locations (1):
- Yale Comprehensive Cancer Center, New Haven, Connecticut, United States